CLINICAL TRIAL: NCT06545799
Title: Construction of a Cohort for Pan-Vascular Disease Among Employees of Taizhou People's Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Jiangsu Taizhou People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY 2024-098-01
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Death; Myocardial Infarction; Stroke
MeSH Terms: conditions — Myocardial Infarction; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — 2 ml of blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

SUMMARY:
1. Participant Recruitment During the annual health check-ups for hospital staff, potential participants are recruited. Those who express interest are provided with a detailed explanation of the study's objectives, content, and procedures, and are required to sign an informed consent form.
2. Screening Phase Medical history is collected, including any previous occurrences of myocardial infarction, ischemic or hemorrhagic stroke, or history of coronary, carotid, or peripheral arterial revascularization.
3. Baseline Data Collection

1. Health Questionnaire Survey: Collect demographic information, medical history, and data on nutrition, physical activity, and smoking habits through a questionnaire.

2. Clinical Assessments: Conduct the following assessments for all enrolled participants:

* High-sensitivity cardiac troponin I and NT-proBNP testing
* Non-invasive arterial stiffness testing
* Measurement of visceral and subcutaneous fat content
* Fundus photography
* Body composition analysis

  4 Regular Follow-Up

Annual follow-up for a total of 10 years. The follow-up includes:

1. . Collection of updated demographic information and medical history, as well as repeated questionnaires on nutrition, physical activity, and smoking habits.
2. . Reassessment of the following items:

   * High-sensitivity cardiac troponin I and NT-proBNP testing
   * Non-invasive arterial stiffness testing
   * Measurement of visceral and subcutaneous fat content
   * Fundus photography
   * Body composition analysis

     5 Outcome Evaluation

1）. Primary Outcomes: Cardiovascular mortality, non-fatal myocardial infarction, or non-fatal stroke events.

2）. Secondary Outcomes: All vascular events, changes in cardiovascular biomarkers, and degree of arterial stiffness.

ELIGIBILITY:
Inclusion Criteria:

1. Employed or retired individuals aged 45 years or older;
2. Willing to sign an informed consent form and voluntarily participate in health examinations and related data collection.

Exclusion Criteria:

1. History of myocardial infarction, ischemic or hemorrhagic stroke, or revascularization of coronary, carotid, or peripheral arteries;
2. Employees with severe psychological disorders who are unable to cooperate with the study;
3. Pregnant or breastfeeding women.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Each year, during the annual health check-ups for hospital staff, potential participants are recruited. Those who express interest are provided with a detailed explanation of the study's objectives, content, and procedures, and are required to sign an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2034-09-01 (Estimated); Study Completion 2034-09-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular death, non-fatal myocardial infarction, or non-fatal stroke events | September 2024 to August 2034
  Cardiovascular death: Death from heart or blood vessel diseases.
  Non-fatal myocardial infarction: Heart attack that does not result in death.
  Non-fatal stroke events: Stroke incidents that do not result in death.

IPD SHARING:
Plan to Share IPD: No